CLINICAL TRIAL: NCT07267117
Title: Cohort Observing Mechanisms, Progression and Sequelae of Valvular Heart Disease (VALVE-COMPASS)
Brief Title: Cohort Observing Mechanisms, Progression and Sequelae of Valvular Heart Disease
Acronym: VALVE-COMPASS
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Army Medical Center of PLA (Other Government); Huaxi Hospital (Other); Fuwai Yunnan Cardiovascular Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Second Xiangya Hospital of Central South University (Other); Xiangya Hospital of Central South University (Other); The General Hospital of Northern Theater Command (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Fujian Provincial Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); The Affiliated Hospital of Qingdao University (Other); Renmin Hospital of Wuhan University (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0528
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-06

CONDITIONS: Heart Valve Disease; Mitral Valve (MV) Regurgitation; Mitral Valve Disease; Mitral Valve Stenosis; Aortic Valve Disease; Aortic Valve Stenosis; Tricuspid Valve Disease; Tricuspid Valve Regurgitation; Aortic Valve Regurgitation; Pulmonary Valve Disease; Transcatheter Valve Replacement; Transcatheter Aortic Valve Replacement (TAVR); Transcatheter Pulmonary Valve Replacement (TPVR); Transcatheter Edge-to-edge Repair
Keywords: Heart Valve Disease Progression; Heart Valve disease sequelae
MeSH Terms: conditions — Heart Valve Diseases; Gastroesophageal Reflux; Mitral Valve Stenosis; Aortic Valve Disease; Aortic Valve Stenosis; Tricuspid Valve Insufficiency; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The patient's blood sample is kept in a suitable way, centrifuged and aliquoted, etc., and stored in a -80° freezer。
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate and predict the progression of moderate cardiac valve stenosis and regurgitation using clinical, biological, echocardiographic, computed tomography (CT), and magnetic resonance imaging (MRI) data. Additionally, the study aims to analyze the potential impact of device-based interventions, pharmacological therapy, and lifestyle modifications on disease progression.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study designed to investigate the disease progression, medication and surgical intervention patterns, outcomes, and influencing factors in patients with moderate or greater cardiac valve stenosis and Grade II or higher cardiac valve regurgitation. The study population includes patients diagnosed at 15 major medical institutions in China, including the Second Affiliated Hospital of Zhejiang University School of Medicine and West China Hospital of Sichuan University. The severity of valvular heart disease is determined according to a standardized dataset (JACC Adv. 2025 Apr) developed by a joint task force comprising multiple international societies.

Currently, there is a lack of clear consensus regarding the management of patients with moderate valvular stenosis and regurgitation, and their subsequent disease progression remains poorly understood. Notably, the time span for progression from moderate to severe valvular heart disease can vary from 1 to 10 years, and monitoring and early warning mechanisms for potential early markers indicating disease deterioration are currently underdeveloped. Furthermore, patients with severe valvular heart disease may experience different outcomes following various device implantations, and the associated risk factors require further clarification.

The objective of this study is to identify all clinical, biological, echocardiographic, and imaging parameters that may increase the risk of disease progression or adverse outcomes through a prospective observational cohort design. The confirmation of these parameters will guide future research in developing pharmacological and interventional treatment strategies to reduce mortality associated with this disease. Patients enrolled in this study will undergo annual outpatient follow-up visits after diagnosis, which will include electrocardiography, echocardiography, blood analysis, and contrast-enhanced CT scans. Through these comprehensive monitoring methods, we aim to accurately assess changes in patients' conditions and provide a scientific basis for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Be willing and able to provide informed consent to participate in the study;
* Patients with heart valve disease diagnosed by echocardiography who meet one of the following criteria:

  1. Grade II or higher Aortic valve regurgitation: regurgitant jet width >3 mm, jet width / LVOT diameter ≥25%, jet cross-sectional area/LVOT cross-sectional area ≥5%, effective regurgitant orifice area (EROA) ≥0.1 cm², regurgitant volume per beat (R Vol)≥30 ml, or regurgitant fraction (RF) ≥30%.
  2. Moderate or higher aortic valve stenosis: peak velocity ≥3.0 m/s, Mean gradient ≥20 mm Hg, aortic valve area ≤1.5 cm², Indexed aortic valve area ≤0.85 cm²/m², or velocity ratio ≤0.50.
  3. Grade II or higher mitral valve regurgitation: regurgitant jet width ≥3 mm, regurgitant volume per beat ≥30 ml, regurgitant jet area/left atrial area >30%, or effective regurgitant orifice area (EROA) ≥0.2 cm².
  4. Moderate or higher valve stenosis: valve area (specific finding) ≤1.5 cm², or mean gradient (supportive finding) ≥10.0 mmHg.
  5. Grade II or higher tricuspid valve regurgitation: regurgitant jet width ≥3 mm, proximal isovelocity surface area ≥6 mm, effective regurgitant orifice area (EROA) ≥0.2 cm², or regurgitant volume per beat ≥30 ml.
  6. Significant tricuspid valve stenosis: mean pressure gradient ≥5.0 mmHg, inflow time-velocity integral >60 cm, T1/2 ≥190 ms, or valve area ≤1.0 cm².
  7. Grade II or higher pulmonary valve regurgitation: regurgitant jet width >3 mm, regurgitant volume per beat ≥30 ml, regurgitant fraction ≥30%, or effective regurgitant orifice area (EROA) ≥0.1 cm².
  8. Moderate or higher Pulmonary valve stenosis: pulmonary valve transvalvular pressure gradient ≥40 mmHg, right ventricular systolic pressure ≥60 mmHg, or pulmonary valve opening <1.5 cm².

Exclusion Criteria:

* Patients who are unwilling to accept registration and follow-up;
* Patients who cannot cooperate with information collection and follow-up due to mental illness or other conditions;
* Patients whose life expectancy is less than 12 months due to non-cardiac diseases (such as cancer, liver disease, kidney disease, or end-stage lung disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective observational cohort study designed to investigate the disease progression, medication and surgical intervention patterns, outcomes, and influencing factors in patients with moderate or greater cardiac valve stenosis and Grade II or higher cardiac valve regurgitation. The study population includes patients diagnosed at 15 major medical institutions in China, including the Second Affiliated Hospital of Zhejiang University School of Medicine and West China Hospital of Sichuan University. The severity of valvular heart disease is determined according to a standardized dataset (JACC Adv. 2025 Apr) developed by a joint task force comprising multiple international societies.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 1-year, 2-year, 3-year, 4-year, and 5-year at follow-up
Heart valve replacement or repair | 1-year, 2-year, 3-year, 4-year, and 5-year at follow-up
  Surgical Heart Valve Replacement/Repair or Transcatheter Aortic Valve Replacement/Repair
Stroke | 1-year, 2-year, 3-year, 4-year, and 5-year at follow-up
  Episode of ischemic stroke or hemorrhagic stroke in the internal carotid artery territory defined on CT scan or MRI brain.
Re-hospitalization related to cardiovascular disease | 1-year, 2-year, 3-year, 4-year, and 5-year at follow-up
  Requires rehospitalization due to cardiovascular diseases such as coronary atherosclerotic heart disease, heart failure, arrhythmia, pulmonary embolism, aortic disease, and hypertension.

SECONDARY OUTCOMES:
Progression of valve stenosis or regurgitation | 1-year, 2-year, 3-year, 4-year, and 5-year at follow-up
  Progression from moderate valvular stenosis to severe stenosis, or from grade II valvular regurgitation to more severe regurgitation, as defined by the echocardiographic examination.
Ventricular remodeling and deterioration of cardiac function | 1-year, 2-year, 3-year, 4-year, and 5-year at follow-up
  Changes in indicators such as LVEF, LVEDD, or anteroposterior diameter of the atria as defined by echocardiography
Changes in quality of life and symptoms | 1-year, 2-year, 3-year, 4-year, and 5-year at follow-up
  NYHA functional class, six-minute walk distance, or newly developed or worsening typical symptoms
Newly Emerging Cardiovascular Disease and Complications | 1-year, 2-year, 3-year, 4-year, and 5-year at follow-up
  Such as newly onset arrhythmic events (including atrial fibrillation/flutter, conduction block, sick sinus syndrome, etc.), non-hospitalized heart failure-related events, bleeding events, thrombotic events, hypertensive emergencies, and symptoms related to myocardial ischemia.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Fujian Provincial Hospital, Affiliated to Fuzhou University, Fuzhou, Fujian
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The First Affiliated Hospital of Air Force Medicial University, Xi'an, Shaanxi
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Huaxi Hospital, Chengdu, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan
  - Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing
  - Navy General Hospital, Beijing, Beijing
  - Army Medical Center of PLA, Chongqing
  - Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lansac E, Veen KM, Joseph A, Blancarte Jaber P, Sossi F, Das-Gupta Z, Aktaa S, Sadaba JR, Thourani VH, Dahle G, Szeto WY, Bakaeen F, Aikawa E, Schoen FJ, Girdauskas E, Almeida A, Zuckermann A, Meuris B, Stott J, Kluin J, Meel R, Woan W, Colgan D, Jneid H, Balkhy H, Szerlip M, Preventza O, Shah P, Rigolin VH, Medica S, Holmes P, Sitges M, Pibarot P, Donal E, Hahn RT, Takkenberg JJM. The First International Consortium for Health Outcomes Measurement (ICHOM) Standard Dataset for Reporting Outcomes in Heart Valve Disease: Moving From Device- to Patient-Centered Outcomes: Developed by a multisociety taskforce coordinated by the Heart Valve Society (HVS) including the American Heart Association (AHA), the American College of Cardiology (ACC), the European Association for Cardio-Thoracic Surgery (EACTS), the European Society of Cardiology (ESC), The Society of Thoracic Surgeons (STS), the Australian & New Zealand Society of Cardiac & Thoracic Surgeons (ANZSCTS), the International Society for Applied Cardiovascular Biology (ISACB), the International Society for Minimally Invasive Cardiothoracic Surgery (ISMICS), the South African Heart Association (SHA), Heart Valve Voice, and Global Heart Hub. JACC Adv. 2025 Apr;4(4):101059. doi: 10.1016/j.jacadv.2024.101059. Epub 2025 Feb 17. PMID 39966045